CLINICAL TRIAL: NCT00695305
Title: A Multicenter, Randomized, 12 Week, Double-blind, Placebo-controlled, Parallel-group, Phase IIa Study Using 18F Fluorodeoxyglucose (FDG)-PET to Measure the Effects of Rilapladib on Macrophage Activity in Subjects With Atherosclerosis
Brief Title: An Imaging Study in Patients With Atherosclerosis Taking Rilapladib or Placebo for 12 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP2105521
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: rilapladib,; Lp-PLA2,; atherosclerosis; SB-659032,; FDG-PET,
MeSH Terms: conditions — Atherosclerosis | interventions — rilapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo to match
  Interventions: Drug: placebo
- rilapladib (Active Comparator): 250 mg/day
  Interventions: Drug: rilapladib; Other: 18F Fluorodeoxylucose (FDG)-PET

INTERVENTIONS:
Drug: rilapladib — 250 mg oral dose once daily
  Other Names: SB-659032
  Arms: rilapladib
Drug: placebo — placebo
  Arms: placebo
Other: 18F Fluorodeoxylucose (FDG)-PET — FDG-PET
  Other Names: FDG marker
  Arms: rilapladib

SUMMARY:
A study in patients with atherosclerosis to assess safety, effect and PK of rilapladib vs. placebo over 12 weeks of dosing.

DETAILED DESCRIPTION:
Study LP2105521 is a randomized, double-blind, placebo-controlled, parallel-group study to examine the safety, tolerability, and effects of rilapladib on plasma Lp-PLA2 activity, plaque inflammation, and PAF (if feasible). Subjects will receive placebo or rilapladib once daily for 12 weeks. The study will be conducted in subjects with established atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent and able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Male or female, aged 50 to 80 years inclusive, at screening.
* Females must be of non-childbearing potential
* Body weight ≥ 50 kg and BMI within the range 19-35 kg/m2
* Documented atherosclerotic vascular disease (e.g. prior MI, prior revascularization, peripheral arterial disease, carotid disease, or cerebrovascular disease) and clinically stable for at least 6 months
* If diabetic, have well controlled diabetes, defined for the purpose of this study as HbA1c ≤8% or FPG ≤200 mg/dL
* Evidence of plaque inflammation [carotid artery or ascending aorta plaque inflammation defined as a tissue to background ratio (TBR) ≥ 1.6]
* On a stable dose of a statin for 3 months prior to screening with no evidence of statin intolerance

Exclusion Criteria:

* Recent (i.e., <6 months from Screening Visit) CV event defined as ST-elevation MI or non-ST-elevation MI, confirmed by cardiac enzyme elevation and ECG changes, coronary revascularization (PCI or CABG), stroke of any etiology, resuscitated sudden death, prior carotid surgery or stenting procedure
* Evidence of clinical instability or abnormal clinical laboratory findings prior to randomization that, in the opinion of the Investigator, makes the subject unsuitable for the study.
* Exposure to substantial radiation within the past 12 months
* Planned cardiac surgery (e.g., CABG, valve repair or replacement, or aneurysmectomy), PCI or major non-cardiac surgery within the study period
* Current inadequately controlled hypertension (blood pressure ≥160 mmHg systolic or ≥100 mmHg diastolic) on a stable dose of anti-hypertensive medication
* Diabetics taking injectable insulin at screening
* Serum triglycerides >400 mg/dL, LDLc >130 mg/dL
* Recent (<1 month) or ongoing acute infection.
* History of chronic inflammatory disease
* Recently received (<1 month) or currently receiving oral or injectable corticosteroids, or regular use of nasal, inhaled or topical corticosteroids.
* Subjects who will commence, or who are likely to commence regular treatment with oral, non-steroidal anti-inflammatory drugs (NSAIDs) from screening until study completion
* Currently receiving oral or injectable potent CYP3A4 inhibitor(s)
* History of chronic viral hepatitis or other chronic hepatic disorders; or ALT or AST >1.5 x ULN, or alkaline phosphatase or total bilirubin >1.5 x ULN of laboratory reference range at Screen
* Renal impairment with serum creatinine >2.0 mg/dl or history of kidney transplant or status post nephrectomy.
* History of myopathy or inflammatory muscle disease, or elevated total CPK at screening
* History of severe heart failure defined as NYHA class III or IV or those with known severe left ventricular dysfunction (ejection fraction<30%) regardless of symptomatic status
* History of adult asthma (or reactive airway disease) manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s)
* History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions or severe allergic responses
* History of malignancy within the past 2 years.
* A history of glaucoma or any other findings in the baseline eye exam
* Current life-threatening condition other than vascular disease that may prevent a subject from completing the study
* QTc interval ≥450msec at screening or ≥480 msec for subjects with bundle branch block
* History of drug abuse within the past 6 months
* Previous exposure to rilapladib.
* Contraindication to MRI scanning
* Use of an investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication
* Any other subject the Investigator deems unsuitable for the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety from AE reporting, vital signs, clinical labs, ECGs, slit lamp eye exams and electron microscopy of peripheral blood lymphocytes. | 12 weeks
LP-PLA2 activity; | 12 weeks
changes in mean standard values of 18 FDG uptake as assessed by PET and MRI imaging | 12 weeks

SECONDARY OUTCOMES:
Estimation of PK parameters (such as: apparent volume of distribution, apparent clearance, etc.) of rilapladib and their associated variability, appropriate to the final model | 12 weeks
Estimation of PK/PD parameters (such as: IC50, Eo) and their associated variability, appropriate to the final model | 12 weeks
24 hour ambulatory blood pressure monitoring | 12 weeks
PAF levels in human plasma as feasible | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Linden, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LP2105521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register